CLINICAL TRIAL: NCT00943254
Title: Metabolic Syndrome: Impact of Receiving the Diagnosis and Education Intervention on Cardiovascular Risk Factor Modification and Willingness to Change
Brief Title: Metabolic Syndrome Diagnosis and Education Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Randal J Thomas, MD, Mayo Clinic- Rohester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-006106
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Metabolic Cardiovascular Syndrome
Keywords: Metabolic Cardiovascular Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Arm 1 (Experimental): Patients randomized to this arm receive the diagnosis of "metabolic syndrome" and subsequent education using paper-based and DVD materials
  Interventions: Other: High-Tech Education
- Arm 2 (Experimental): Patients in this arm receive the diagnosis of "metabolic syndrome" and subsequent education using paper-based material
  Interventions: Other: Low-Tech Education
- Arm 3 (No Intervention): Patients randomized to control receive the diagnosis of individual cardiovascular risk factors with paper-based educational material

INTERVENTIONS:
Other: High-Tech Education — Patients will be told that they have the metabolic syndrome and will subsequently watch two 10-minute videos on the metabolic syndrome and on getting started with exercise. They also receive all the paper-based educational material as in arm 2
  Arms: Arm 1
Other: Low-Tech Education — Patients will be told that they have the metabolic syndrome and will subsequently receive paper-based educational material on the metabolic syndrome,pre-diabetes, and hypertension. They also receive pamphlets on dietary management of high cholesterol and triglycerides, and the importance of exercise and weight loss.
  Arms: Arm 2

SUMMARY:
This study is being done to gain knowledge on how effective different approaches of providing a diagnosis and varying educational tools that include DVDs and multimedia or printed instruction sheets on your readiness to increase the subject's level of exercise, lose more weight, eat a healthier diet; and to assess the subject's awareness of their risk of heart disease and their readiness to participate in a comprehensive lifestyle modification program.

ELIGIBILITY:
Inclusion Criteria:

Any 3 of the following 5:

1. History of hypertension or either systolic blood pressure >125 or diastolic blood pressure >85 mmHg or documented history and receiving treatment for it
2. Abdominal circumference ≥40 inches in men or ≥35 inches in women
3. Fasting triglycerides ≥ 150mg/dL or receiving treatment for it
4. Fasting blood glucose ≥ 100mg/dL but <126mg/dL
5. HDL cholesterol <40mg/dL in men or <50mg/dL in women or receiving treatment for it

Exclusion Criteria:

1. Documented diagnosis of metabolic syndrome in the clinical record, if previously seen at Mayo.
2. History of coronary artery disease
3. Diabetes mellitus, or using an oral hypoglycemic pill for glucose intolerance
4. Congestive heart failure
5. Familial hypercholesterolemia including familial hypertriglyceridemia,
6. Fasting LDL-cholesterol >160 mg/dL
7. Fasting triglycerides > 390 mg/dL
8. Have systolic blood pressure >160 and diastolic blood pressure >100mg/dL
9. History of hypertension with changes in their blood pressure medicines within the last 60 days before enrollment.
10. History of dyslipidemia and changes on their lipid lowering agents such as statins, ezetimibe, fibrates or niacin within the last 60 days before enrollment.
11. Secondary causes of obesity such as hypothyroidism, Cushing syndrome, or eating disorders
12. Pregnant women or women planning to get pregnant during the duration of the study
13. Advanced liver disease
14. Renal insufficiency
15. Having any other major chronic medical condition
16. Unable to do their basic chores at home due to musculoskeletal limitations or other factors affecting their functional status.
17. Physical activity of more than 60 minutes per week of moderate to intense exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Lifestyle Change: Readiness to Exercise, level of physical activity | 6 weeks
Stages of Change for Exercise and for Fruits and vegetables | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Randal J Thomas, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Jumean MF, Korenfeld Y, Somers VK, Vickers KS, Thomas RJ, Lopez-Jimenez F. Impact of diagnosing metabolic syndrome on risk perception. Am J Health Behav. 2012 Jul;36(4):522-32. doi: 10.5993/AJHB.36.4.9. PMID 22488402